CLINICAL TRIAL: NCT03709693
Title: Sternal Rigid Fixation: Evaluation of Clinical Outcomes Using Real-World Evidence
Brief Title: Clinical Outcomes in Patients Treated With SternaLock Blu
Acronym: SECURE
Status: Terminated | Type: Observational
Why Stopped: COVID 19 Pandemic
Sponsor: Zimmer Biomet (Industry)
Responsible Party: Sponsor
Other Study IDs: 0518
Record Dates: First submitted 2018-10-16; First posted 2018-10-17 (Actual); Last update posted 2021-07-23 (Actual); Status verified 2021-07

CONDITIONS: Cardiac Surgical Procedures; Coronary Artery Disease; Heart Valve Diseases
Keywords: sternotomy; rigid fixation; sternal fixation; sternal plating
MeSH Terms: conditions — Coronary Artery Disease; Heart Valve Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 90 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- SternaLock Blu: All patients will receive SternaLock Blu for closure of full mid-line sternotomy.
  Interventions: Device: SternaLock Blu

INTERVENTIONS:
Device: SternaLock Blu — Sternal closure will be accomplished using SternaLock Blu plates and screws in combination with single-wire method of sternal reduction.

SUMMARY:
The primary objective of this study is to evaluate the rate of deep sternal wound infection at 30 days post-operative following a full median sternotomy in patients treated with SternaLock Blu for rigid sternal fixation. This study will also provide evidence of the clinical performance of SternaLock Blu for up to 90 days using real world evidence methodology. Sternal complications will be reported through 90 days follow up.

DETAILED DESCRIPTION:
The primary endpoint for this study is the rate of deep sternal wound infection (DSWI) at 30 days post-operative, following a midline sternotomy closed with SternaLock Blu. DSWI is defined as deep infection involving muscle, bone, and/ or mediastinum requiring operative intervention and has all of the following conditions:

1. Wound opened with excision of tissue or re-exploration of mediastinum
2. Positive culture unless patient on antibiotics at the time of culture or no culture obtained
3. Treatment with antibiotics beyond perioperative prophylaxis

Post-operative sternal wound complications occurring within 90 days post-operative.

Outcomes will be reported up to 90 days after surgery, including data on adverse events associated with the use of SternaLock Blu Sternal Closure System from the moment of implantation to the end-of-study.

ELIGIBILITY:
Inclusion Criteria:

1. ≥ 18 years of age, no upper limit
2. Undergoing a full standard midline sternotomy as part of an elective or urgent cardiac surgical procedure [i.e., coronary artery bypass graft (CABG) and/ or valve replacement along with other cardiac surgical procedures] and closed with the SternaLock Blu Sternal Closure System
3. Willing and able to return for follow-up

   Exclusion Criteria:

   Preoperative
4. Emergent or salvage cardiac acuity i.e., patients undergoing cardiopulmonary resuscitation en-route to the operating room or prior to induction of anesthesia
5. Any contraindication listed in the SternaLock Blu instructions for use (IFU/ Appendix 3) (active infection, foreign body sensitivity, or mental/ neurologic conditions who are unwilling or incapable of following post-operative care instructions) Operative
6. Delayed sternal closure required for any reason
7. Intra-operative conditions that, in the opinion of the operating surgeon, would preclude the use of rigid plate fixation, i.e.: insufficient quantity of sternal bone or compressible sternum indicating poor bone quality, as assessed by the operating surgeon using his or her professional judgment at the time of closure
8. Use of bone wax between the sternal halves
9. Intraoperative death prior to device placement

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 2000 subjects total (+/- 20) from up to 20 sites
Sampling Method: Probability Sample
Enrollment: 156 (Actual)
Dates: Start 2019-05-14 (Actual); Primary Completion 2020-05-13 (Actual); Study Completion 2020-05-13 (Actual)

PRIMARY OUTCOMES:
Deep Sternal Wound Infection Rate | at 30 days post operatively up to 90 days
  DSWI is defined as deep infection involving muscle, bone, and/ or mediastinum requiring operative intervention and has all of the following conditions:
  1. Wound opened with excision of tissue (I&D) or re-exploration of mediastinum
  2. Positive culture unless patient on antibiotics at the time of culture or no culture obtained
  3. Treatment with antibiotics beyond perioperative prophylaxis

CONTACTS AND LOCATIONS:
Overall Officials: Keith Allen, MD, Principal Investigator — St. Luke's Hospital; Marc Gerdisch, MD, Principal Investigator — St Franciscan Health
Locations (4):
- United States (4):
  - St. Franciscan Health, Indianapolis, Indiana
  - Saint Luke's Hospital of Kansas City, Kansas City, Missouri
  - Cardiovascular Surgery Clinic, PLLC, Memphis, Tennessee
  - University of Virginia, Charlottesville, Virginia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Adams J, Schmid J, Parker RD, Coast JR, Cheng D, Killian AD, McCray S, Strauss D, McLeroy Dejong S, Berbarie R. Comparison of force exerted on the sternum during a sneeze versus during low-, moderate-, and high-intensity bench press resistance exercise with and without the valsalva maneuver in healthy volunteers. Am J Cardiol. 2014 Mar 15;113(6):1045-8. doi: 10.1016/j.amjcard.2013.11.064. Epub 2013 Dec 25. PMID 24440333
- [Background] O'Brien SM, Shahian DM, Filardo G, Ferraris VA, Haan CK, Rich JB, Normand SL, DeLong ER, Shewan CM, Dokholyan RS, Peterson ED, Edwards FH, Anderson RP; Society of Thoracic Surgeons Quality Measurement Task Force. The Society of Thoracic Surgeons 2008 cardiac surgery risk models: part 2--isolated valve surgery. Ann Thorac Surg. 2009 Jul;88(1 Suppl):S23-42. doi: 10.1016/j.athoracsur.2009.05.056. PMID 19559823
- [Background] Sharma R, Puri D, Panigrahi BP, Virdi IS. A modified parasternal wire technique for prevention and treatment of sternal dehiscence. Ann Thorac Surg. 2004 Jan;77(1):210-3. doi: 10.1016/s0003-4975(03)01339-0. PMID 14726063
- [Background] Shifrin DA, Sohn SM, Stouffer CW, Hooker RL, Renucci JD. Sternal salvage with rigid fixation in the setting of a massive mediastinal aortic pseudoaneurysm: a case report and review of the literature. J Plast Reconstr Aesthet Surg. 2008 Oct;61(10):e17-20. doi: 10.1016/j.bjps.2007.09.022. Epub 2007 Nov 26. PMID 18033747
- [Background] Song DH, Lohman RF, Renucci JD, Jeevanandam V, Raman J. Primary sternal plating in high-risk patients prevents mediastinitis. Eur J Cardiothorac Surg. 2004 Aug;26(2):367-72. doi: 10.1016/j.ejcts.2004.04.038. PMID 15296898
- [Background] RESTORE (2012).
- [Background] Quality M (2012).
- [Background] Neaman KC, Blount AL, Kim JA, Renucci JD, Hooker RL. Prophylactic sternal plating with pectoralis advancement flaps after sternotomy in patients with a history of chest irradiation. Interact Cardiovasc Thorac Surg. 2011 Mar;12(3):355-8. doi: 10.1510/icvts.2010.247262. Epub 2010 Dec 7. PMID 21138917
- [Background] Gorlitzer M, Wagner F, Pfeiffer S, Folkmann S, Meinhart J, Fischlein T, Reichenspurner H, Grabenwoger M. A prospective randomized multicenter trial shows improvement of sternum related complications in cardiac surgery with the Posthorax support vest. Interact Cardiovasc Thorac Surg. 2010 May;10(5):714-8. doi: 10.1510/icvts.2009.223305. Epub 2010 Jan 26. PMID 20103509
- [Background] Fedak PW, Kieser TM, Maitland AM, Holland M, Kasatkin A, Leblanc P, Kim JK, King KM. Adhesive-enhanced sternal closure to improve postoperative functional recovery: a pilot, randomized controlled trial. Ann Thorac Surg. 2011 Oct;92(4):1444-50. doi: 10.1016/j.athoracsur.2011.05.014. PMID 21958795
- [Background] Dickie SR, Dorafshar AH, Song DH. Definitive closure of the infected median sternotomy wound: a treatment algorithm utilizing vacuum-assisted closure followed by rigid plate fixation. Ann Plast Surg. 2006 Jun;56(6):680-5. doi: 10.1097/01.sap.0000202825.41069.c3. PMID 16721085
- [Background] Clopper CJ (1934) The use of confidcence or fiducial limits illustrated in the case of the binomial. Biometrika 26(4): 404-413.
- [Background] CCS
- [Result] Casha AR, Yang L, Kay PH, Saleh M, Cooper GJ. A biomechanical study of median sternotomy closure techniques. Eur J Cardiothorac Surg. 1999 Mar;15(3):365-9. doi: 10.1016/s1010-7940(99)00014-7. PMID 10333037
- [Result] Claes L, Augat P, Suger G, Wilke HJ. Influence of size and stability of the osteotomy gap on the success of fracture healing. J Orthop Res. 1997 Jul;15(4):577-84. doi: 10.1002/jor.1100150414. PMID 9379268
- [Result] D'Agostino RS, Jacobs JP, Badhwar V, Paone G, Rankin JS, Han JM, McDonald D, Shahian DM. The Society of Thoracic Surgeons Adult Cardiac Surgery Database: 2016 Update on Outcomes and Quality. Ann Thorac Surg. 2016 Jan;101(1):24-32. doi: 10.1016/j.athoracsur.2015.11.032. Epub 2015 Nov 24. PMID 26616408
- [Result] Gottlieb LJ, Pielet RW, Karp RB, Krieger LM, Smith DJ Jr, Deeb GM. Rigid internal fixation of the sternum in postoperative mediastinitis. Arch Surg. 1994 May;129(5):489-93. doi: 10.1001/archsurg.1994.01420290035005. PMID 8185470
- [Result] Lahtinen P, Kokki H, Hynynen M. Pain after cardiac surgery: a prospective cohort study of 1-year incidence and intensity. Anesthesiology. 2006 Oct;105(4):794-800. doi: 10.1097/00000542-200610000-00026. PMID 17006079
- [Result] Losanoff JE, Collier AD, Wagner-Mann CC, Richman BW, Huff H, Hsieh Fh, Diaz-Arias A, Jones JW. Biomechanical comparison of median sternotomy closures. Ann Thorac Surg. 2004 Jan;77(1):203-9. doi: 10.1016/s0003-4975(03)01468-1. PMID 14726062
- [Result] Meyerson J, Thelin S, Gordh T, Karlsten R. The incidence of chronic post-sternotomy pain after cardiac surgery--a prospective study. Acta Anaesthesiol Scand. 2001 Sep;45(8):940-4. doi: 10.1034/j.1399-6576.2001.450804.x. PMID 11576043
- [Result] Pai S, Gunja NJ, Dupak EL, McMahon NL, Coburn JC, Lalikos JF, Dunn RM, Francalancia N, Pins GD, Billiar KL. A mechanical study of rigid plate configurations for sternal fixation. Ann Biomed Eng. 2007 May;35(5):808-16. doi: 10.1007/s10439-007-9272-3. Epub 2007 Mar 22. PMID 17377844
- [Result] Raman J, Straus D, Song DH. Rigid plate fixation of the sternum. Ann Thorac Surg. 2007 Sep;84(3):1056-8. doi: 10.1016/j.athoracsur.2006.11.045. PMID 17720442
- [Result] Sargent LA, Seyfer AE, Hollinger J, Hinson RM, Graeber GM. The healing sternum: a comparison of osseous healing with wire versus rigid fixation. Ann Thorac Surg. 1991 Sep;52(3):490-4. doi: 10.1016/0003-4975(91)90910-i. PMID 1898136
- [Result] Vassileva CM, Aranki S, Brennan JM, Kaneko T, He M, Gammie JS, Suri RM, Thourani VH, Hazelrigg S, McCarthy P. Evaluation of The Society of Thoracic Surgeons Online Risk Calculator for Assessment of Risk in Patients Presenting for Aortic Valve Replacement After Prior Coronary Artery Bypass Graft: An Analysis Using the STS Adult Cardiac Surgery Database. Ann Thorac Surg. 2015 Dec;100(6):2109-15; discussion 2115-6. doi: 10.1016/j.athoracsur.2015.04.149. Epub 2015 Jul 30. PMID 26233279
- [Result] STS
- [Result] Snyder CW, Graham LA, Byers RE, Holman WL. Primary sternal plating to prevent sternal wound complications after cardiac surgery: early experience and patterns of failure. Interact Cardiovasc Thorac Surg. 2009 Nov;9(5):763-6. doi: 10.1510/icvts.2009.214023. Epub 2009 Aug 26. PMID 19710069
- [Result] Schimmer C, Sommer SP, Bensch M, Bohrer T, Aleksic I, Leyh R. Sternal closure techniques and postoperative sternal wound complications in elderly patients. Eur J Cardiothorac Surg. 2008 Jul;34(1):132-8. doi: 10.1016/j.ejcts.2008.04.006. Epub 2008 May 9. PMID 18468447
- [Result] Schimmer C, Reents W, Berneder S, Eigel P, Sezer O, Scheld H, Sahraoui K, Gansera B, Deppert O, Rubio A, Feyrer R, Sauer C, Elert O, Leyh R. Prevention of sternal dehiscence and infection in high-risk patients: a prospective randomized multicenter trial. Ann Thorac Surg. 2008 Dec;86(6):1897-904. doi: 10.1016/j.athoracsur.2008.08.071. PMID 19022005
- [Result] Raman J, Song DH, Bolotin G, Jeevanandam V. Sternal closure with titanium plate fixation--a paradigm shift in preventing mediastinitis. Interact Cardiovasc Thorac Surg. 2006 Aug;5(4):336-9. doi: 10.1510/icvts.2005.121863. Epub 2006 Apr 25. PMID 17670585
- [Result] NYHA
- [Result] Losanoff JE, Basson MD, Gruber SA, Huff H, Hsieh FH. Single wire versus double wire loops for median sternotomy closure: experimental biomechanical study using a human cadaveric model. Ann Thorac Surg. 2007 Oct;84(4):1288-93. doi: 10.1016/j.athoracsur.2007.05.023. PMID 17888985
- [Result] Lee JC, Raman J, Song DH. Primary sternal closure with titanium plate fixation: plastic surgery effecting a paradigm shift. Plast Reconstr Surg. 2010 Jun;125(6):1720-1724. doi: 10.1097/PRS.0b013e3181d51292. PMID 20517097
- [Result] JULIAN OC, LOPEZ-BELIO M, DYE WS, JAVID H, GROVE WJ. The median sternal incision in intracardiac surgery with extracorporeal circulation; a general evaluation of its use in heart surgery. Surgery. 1957 Oct;42(4):753-61. No abstract available. PMID 13467646
- [Result] Hirose H, Yamane K, Youdelman BA, Bogar L, Diehl JT. Rigid sternal fixation improves postoperative recovery. Open Cardiovasc Med J. 2011;5:148-52. doi: 10.2174/1874192401105010148. Epub 2011 Jul 4. PMID 21760857
- [Result] Collin C, Wade DT, Davies S, Horne V. The Barthel ADL Index: a reliability study. Int Disabil Stud. 1988;10(2):61-3. doi: 10.3109/09638288809164103. PMID 3403500
- [Result] Cohen DJ, Griffin LV. A biomechanical comparison of three sternotomy closure techniques. Ann Thorac Surg. 2002 Feb;73(2):563-8. doi: 10.1016/s0003-4975(01)03389-6. PMID 11845875
- [Result] Chou SS, Sena MJ, Wong MS. Use of SternaLock plating system in acute treatment of unstable traumatic sternal fractures. Ann Thorac Surg. 2011 Feb;91(2):597-9. doi: 10.1016/j.athoracsur.2010.07.083. PMID 21256325
- [Result] Biomet (2012). SternaLock Blu Primary Closure System Brochure. Biomet Microfixation.
- [Result] Bennett-Guerrero E, Phillips-Bute B, Waweru PM, Gaca JG, Spann JC, Milano CA. Pilot study of sternal plating for primary closure of the sternum in cardiac surgical patients. Innovations (Phila). 2011 Nov;6(6):382-8. doi: 10.1097/IMI.0b013e318248fbda. PMID 22436774
- [Result] Atkins, Z. B., & Wolfe, W. G. (2012). Sternal wound complications following cardiac surgery. In Special Topics in Cardiac Surgery. InTech.
- [Result] Allen KB, Thourani VH, Naka Y, Grubb KJ, Grehan J, Patel N, Guy TS, Landolfo K, Gerdisch M, Bonnell M, Cohen DJ. Rigid Plate Fixation Versus Wire Cerclage: Patient-Reported and Economic Outcomes From a Randomized Trial. Ann Thorac Surg. 2018 May;105(5):1344-1350. doi: 10.1016/j.athoracsur.2017.12.011. Epub 2018 Jan 11. PMID 29337126
- [Result] Allen KB, Thourani VH, Naka Y, Grubb KJ, Grehan J, Patel N, Guy TS, Landolfo K, Gerdisch M, Bonnell M, Cohen DJ. Randomized, multicenter trial comparing sternotomy closure with rigid plate fixation to wire cerclage. J Thorac Cardiovasc Surg. 2017 Apr;153(4):888-896.e1. doi: 10.1016/j.jtcvs.2016.10.093. Epub 2016 Nov 17. PMID 27923485